CLINICAL TRIAL: NCT06002789
Title: Safety and Efficacy of PD-1 Monoclonal Antibody With or Without mFOLFOX6 Neoadjuvant Therapy in Patients With Local Advanced Deficient Mismatch Repair/Microsatellite Instability-high Synchronous Multiple Primary Colorectal Cancer (sMPCC)
Brief Title: Safety and Efficacy of PD-1 ± mFOLFOX6 Neoadjuvant Therapy in Local Advanced sMPCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2023073
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Multiple Cancer; Colorectal Cancer
Keywords: Synchronous multiple primary colorectal cancer; PD-1; Neoadjuvant treatment; MSI-H
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: MSI-H/MSS (dMMR/pMMR) mixed sMPCC or all-MSI-H (dMMR) sMPCC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSI-H/MSS (dMMR/pMMR) mixed sMPCC or all-MSI-H (dMMR) sMPCC (Experimental): 1. MSI-H/MSS (dMMR/pMMR) mixed sMPCC: Synchronous multiple primary colorectal cancer consist of MSI/dMMR and MSS/pMMR tumors at the same time
  2. all-MSI-H (dMMR) sMPCC: Synchronous multiple primary colorectal cancer with all MSI/dMMR tumors
  Interventions: Drug: MSI-H/MSS (dMMR/pMMR) mixed sMPCC: combination of mFOLFOX6+PD-1 monoclonal antibody neoadjuvant therapy; Drug: All-MSI-H (dMMR) sMPCC: single-drug PD-1 monoclonal antibody neoadjuvant therapy

INTERVENTIONS:
Drug: MSI-H/MSS (dMMR/pMMR) mixed sMPCC: combination of mFOLFOX6+PD-1 monoclonal antibody neoadjuvant therapy — For MSI-H/MSS (dMMR/pMMR) mixed sMPCC, a combination of neoadjuvant chemotherapy with mFOLFOX6 and immunotherapy with PD-1 monoclonal antibody are applied.
  Other Names: Mixed sMPCC
Drug: All-MSI-H (dMMR) sMPCC: single-drug PD-1 monoclonal antibody neoadjuvant therapy — For all-MSI-H (dMMR) sMPCC, single-drug PD-1 monoclonal antibody immunotherapy is applied.
  Other Names: MSI-H sMPCC

SUMMARY:
At present, radical resection ± preoperative neoadjuvant chemotherapy for colorectal cancer is still the standard comprehensive treatment. In recent years, immunotherapy of PD-1 monoclonal antibody has a significant effect in the second-line/first-line treatment of dMMR/MSI-H advanced colorectal cancer and the neoadjuvant treatment of early colorectal cancer. Synchronous multiple primary colorectal cancer (sMPCC) is a relatively rare type of colorectal cancer (CRC) that refers to the simultaneous occurrence of 2 or more independent primary malignancies in the colon or rectum. The recent large-scale, single-center retrospective study of the investigator showed that compared with single primary colorectal cancer (SPCRC)patients, the incidence of dMMR/MSI-H was significantly higher in sMPCC patients. Besides, a certain proportion of sMPCC patients could both have MSI and MSS tumors at the same time. There is no standard regimen for this patients so far. This study intends to treat the MSI-H/MSS (dMMR/pMMR) mixed sMPCC patients with combination of mFOLFOX6+PD-1 monoclonal antibody neoadjuvant therapy, and treat the all-MSI-H (dMMR) sMPCC patients with single-drug PD-1 monoclonal antibody neoadjuvant therapy. Given the current gaps in the guideline, the investigator intends to take the lead in carrying out this open, multi-center, prospective clinical phase II study. This study might provide a clinical evidence for individual treatment of sMPCC patients, in preserving the functions and organs to the greatest extent.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common malignant tumors in the world. At present, radical resection ± preoperative neoadjuvant chemotherapy for colorectal cancer is still the standard comprehensive treatment recommended by the two major international guidelines of NCCN and ESMO, as well as the Chinese CSCO guidelines. Mismatch repair protein (MMR) expression and microsatellite instability (MSI) status are important factors affecting the efficacy of immunotherapy. In recent years, immunotherapy of PD-1 monoclonal antibody has a significant effect in the second-line/first-line treatment of dMMR/MSI-H advanced colorectal cancer and the neoadjuvant treatment of early colorectal cancer, all of which have shown very good efficacy with great safety and tolerable toxicity.

Synchronous multiple primary colorectal cancer (sMPCC) is a relatively rare type of colorectal cancer (CRC) that refers to the simultaneous occurrence of 2 or more independent primary malignancies in the colon or rectum of the same patient. Since 2000, the annual incidence and mortality of CRC in China have continued to increase, and the incidence of sMPCC has also increased. The overall incidence of sMPCC ranges from 1.1% to 8.1% of CRC patients. The recent large-scale, single-center retrospective study of the investigator showed that among 239 sMPCC patients, the proportions of all-pMMR, all-dMMR, and mixed types (pMMR/dMMR) were 189 (79.1%), 40 (16.7%), and 10 (4.2%), respectively. Compared with single primary colorectal cancer (SPCRC) patients, the incidence of dMMR was significantly higher in sMPCC patients (50/239 vs 872/13037). The results of NGS detection of MSI status were consistent with the results of Immunohistochemistry (IHC), 21.8% (17/78) of sMPCC patients were MSI-H, while the proportion was only 5.3% (5/94) in SPCRC patients. At present, single-drug PD-1 or combined with other immunotherapy has become the first-line treatment for MSI-H SPCRC patients. However, there is no standard regimen for some sMPCC patients who both have MSI-H and MSS lesions. Moreover, there are no studies and reports on the treatment of mFOLFOX6+PD-1 monoclonal antibody in MSI-H/MSS mixed sMPCC and PD-1 monoclonal antibody in all-MSI-H sMPCC.

This study intends to treat the MSI-H/MSS (dMMR/pMMR) mixed sMPCC patients with combination of mFOLFOX6+PD-1 monoclonal antibody neoadjuvant therapy, and treat the all-MSI-H (dMMR) sMPCC patients with single-drug PD-1 monoclonal antibody neoadjuvant therapy. As one of the largest single centers for the diagnosis and treatment of colorectal cancer in China, the Sixth Affiliated Hospital of Sun Yat-sen University has performed nearly 4,000 cases of colorectal cancer surgery per year. Therefore, the investigator intends to take the lead in carrying out this open, multi-center, prospective clinical phase II study in the world. The investigator will give different treatments by the result of microsatellite instability status of all lesions in sMPCC. The pCR rate, incidence of AEs of neoadjuvant therapy, R0 resection rate, down-stage rate, 3 years DFS rate and OS rate are analyzed. This study might provide a clinical evidence for individual treatment of sMPCC patients, in preserving the functions and organs to the greatest extent.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of simultaneous multiple primary colorectal cancer (sMPCC);
2. Tumor biopsy immunohistochemistry of at least one tumor lesion identified dMMR, including the expression loss of one or more of the four proteins MSH1, MSH2, MSH6 and PMS2; or at least one tumor lesion identified MSI-H by polymerase chain reaction or next-generation sequencing technique;
3. Clinical staging T3-4NxM0, with or without positive MRF, with or without positive EMVI;
4. Staging method: all patients undergo chest,abdominal and pelvic enhanced CT, rectal palpation, high resolution MRI examination，positive perienteric lymph node(LN): short diameter ≥10mm LN or LN with typical metastatic shape and MRI character, clinical data should be re-evaluated and judged by center evaluation group when there are contradictory stagings，distant metastasis were excluded by chest and abdominal enhanced CT and pelvic enhanced MRI;
5. No intestinal obstruction symptom，or obstruction relieved after proximal colostomy;
6. No colorectal surgery history;
7. No chemotherapy or radiotherapy history;
8. No biopharmaceutical treatment history(such as monoclonal antibody), immunotherapy(such as anti PD-1antibody, anti PD-L1 antibody, anti PD-L2 antibody or anti CTLA-4), or other research drug treatment;
9. No endocrinotherapy history restriction;
10. informed consent assigned.

Exclusion Criteria:

1. Arrhythmia need anti-arrhythmia treatment(except β-blocking agent or Digoxin), symptomatic coronary heart disease or myocardial ischemia(myocardial infarction within 6 months) or congestive heart-failure (CHF) > NYHA grade II;
2. Severe hypertension not well controlled by drugs;
3. HIV infection history or active phase of chronic Hepatitis B or C(high copies of virus DNA);
4. Active tuberculosis(TB), accepting anti-TB treatment or anti-TB treatment within 1 year before trial screen;
5. Other active clinical severe infection(NCI-CTC AE V5.0);
6. Outside pelvic distant metastasis evidences;
7. Dyscrasia, organ dysfunction;
8. Pelvic or abdominal radiotherapy history;
9. Epilepsy need treatments(Steroid or anti-epilepsy therapy);
10. Other malignant tumor history within 5 years;
11. Over abuse of drugs, medical and psychological or social conditions that might interfere patients or evaluation of the study results;
12. Any active autoimmune disease or autoimmune disease history (including but not restricted: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism, asthma need bronchodilators);
13. Any anti-infection vaccine injection 4 weeks before inclusion;
14. Long-term exposure to immune-suppressor, combination of systemic or topical use of corticosteroids (dose>10mg/day prednisolone or equivalent hormone);
15. Known or suspicious allergy to any study related drugs;
16. Any unstable state might cause damage to the safety and compliance of patients;
17. Pregnant or breast feeding women who has ability to have children while without contraception;
18. Refuse to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 1 year
  pathological complete remission rate

SECONDARY OUTCOMES:
Incidence rate of Grade ≥3 PD-1monoclonal antibody-related adverse events | 1 year
  Incidence rate of participants with Grade ≥3 PD-1monoclonal antibody-related adverse events as assessed by CTCAE v4.0
Incidence rate of Grade ≥3 chemotherapy-related adverse events | 1 year
  Incidence rate of participants with Grade ≥3 chemotherapy-related adverse adverse events as assessed by CTCAE v4.0
R0 resection rate | 1 year
  R0 resection rate in participants treated after mFOLFOX6+Bevacizumab+PD-1monoclonal antibody
Down-stage rate | 1 year
  Down-stage rate of pathological stage after surgery compared with clinical stage before drug treatment
3 years DFS Rate | 3 years
  3 years Disease Free Survival Rate
3 years OS Rate | 3 years
  3 years Overall Survival Rate

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yatsen University, Guangzhou, Guangdong, China